CLINICAL TRIAL: NCT05345353
Title: Weight Development in Children With Severe Obesity After Participation in Two Different Municipal Family-centered Lifestyle Interventions
Brief Title: Childhood Obesity, Lifestyle Interventions and Weight Development
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus Kommune (Other); Randers Municipality, Denmark (Other)
Responsible Party: Principal Investigator, Rasmus Møller Jørgensen, Principal Investigator, Medical Doctor, PhD student at Institute for Clinical Medicin, Health, AU, University of Aarhus
Other Study IDs: 2596
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Pediatric Obesity
Keywords: Lifestyle Intervention; Long term follow-up; Weight developement
MeSH Terms: conditions — Pediatric Obesity | interventions — CD36 Antigens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The Aarhus Protocol, Aarhus municipality:: Children with obesity who participated in a family-centered multicomponent lifestyle intervention - The Aarhus Protocol, Aarhus Municipality
  Interventions: Behavioral: Fat For Fight (FFF), The Aarhus Protocol
- The Randers Protocol, Randers municipality:: children with obesity who participated in a family-centered multicomponent lifestyle Intervention - The Randers Protocol: Randers Municipality
  Interventions: Behavioral: The Children's Obesity Clinic Treatment (TCOCT), The Randers Protocol
- No intervention: Children with obesity who didn't participate in a lifestyle intervention delivered by the municipality.

INTERVENTIONS:
Behavioral: Fat For Fight (FFF), The Aarhus Protocol — A multicomponent family-centered lifestyle intervention which included visits at home and weekly supervised physical activity. Intervention duration - one year maximum
  Groups: The Aarhus Protocol, Aarhus municipality:
Behavioral: The Children's Obesity Clinic Treatment (TCOCT), The Randers Protocol — A multicomponent family-centered lifestyle intervention which included repeatedly visits (up to 8 times / year). Intervention duration - three years maximum
  Groups: The Randers Protocol, Randers municipality:

SUMMARY:
Childhood obesity has been associated with increased risk of both continued excess body weight, development of non-communicable lifestyle diseases and impaired mental health.

Approximately 800 children with obesity were treated with a municipality based family-centered lifestyle intervention in the time period 2010-2020. In the same time period, approximately 2000 children with obesity who did not receive any treatment have been identified.

Our aim is to investigate the efficiency of the two interventions and compare those to children not receiving any treatment. We will use data from both the clinical visits at the municipality health care workers and data from Statistics Denmark.

DETAILED DESCRIPTION:
Childhood obesity often track into adolescence and adulthood resulting in elevated risk of non-communicable lifestyle diseases (e.g. type 2 diabetes). Furthermore, children with obesity are also at risk for impaired mental health (i.e. reduced cognitive function and happiness) and psychological ill-being (i.e. depression, anxiety) compared to their lean peers. Finding methods to efficiently, and in a sustainable way, to treat childhood overweight or obesity has not yet been described.

The aim of this study is therefore to investigate the long term effects of two well established lifestyle interventions on weight development (BMI z-score) and to compare socioeconomic parameters between the intervention groups and children who did not received treatment.

The interventions:

The Aarhus protocol: A multicomponent family-centered lifestyle intervention including visits at home and an opportunity for weekly supervised training. The duration of the intervention was a maximum of one year. Data is available from January 2010.

The Randers Protocol: A multicomponent family-centered lifestyle intervention including repeated visits (up to 8 times each year). The duration of the intervention was a maximum of three years. Data is available from January 2014.

The participants:

Inclusion criteria were children aged 4-18 years with obesity (BMI z-score above the 99. percentile for gender and age) living in Aarhus or Randers municipality.

Between 2010-2020, the following children were included in this trial:

* app. 500 children treated with the Aarhus Protocol,
* app. 300 children treated with the Randers Protocol and
* app. 2000 children in Aarhus who did not participate in a lifestyle intervention delivered by the municipality.

The children were examined routinely (a minimum of three times during elementary school) by the school nurse and anthropometrics were collected in NOVAX. NOVAX is a broadly used IT system which stores and delivers data on childhood anthropometrics to the national the database.

Data collection & analyses:

The weight development will be assessed using data from the municipality and data from the NOVAX. Socioeconomic status will be assessed using register data from Statistics Denmark.

Ethics & permissions:

The local committee on health ethics have approved the overall project and data transfer (rec.no 1-45-70-27-2) The project is internally reported to the University of Aarhus (rec no. 2596) The project has achieved approval from The Danish Data Protection Agency and the Principal Investigator has been granted accessed to data from registers from Danish Statistics.

The project has been reported to ClinicalTrials.gov. The researchers have no conflict of interest to declare.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI z-score above the 99. percentile for gender and age)

Exclusion Criteria:

* No Obesity
* Treatment started outside the inclusion period

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with obesity, 4-18 years of age living in Aarhus or Randers municipality between 2010-2020. The children have either received treatment with a community based lifestyle intervention or received no treatment.
Sampling Method: Non-Probability Sample
Enrollment: 2898 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Weight development as assessed by BMI z-score: | The Aarhus Protocol: 1st of January 2010 to 1st of June 2020. The Randers Protocol: 1st of January 2014 to 1st of June 2020. No Intervention: 1st of January 2010 to 1st of June 2020.
  The weight development will be assessed in all children, who participated in one of two different lifestyle interventions compared to children with no intervention. The weight development will also be assessed in subgroups of the cohort, such as children who did not completed the intervention or who not did participation in the exercise part of the interventions.

SECONDARY OUTCOMES:
Socioeconomic differences, subgroup differences | Socioeconomic data will be assessed at the time of inclusion for each subject.
  socioeconomic differences between children in the interventions, different subgroups and children with no intervention.
  Socioeconomic data will be collected from Danish Statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
participant data (IPD) will be available on reasonable request